CLINICAL TRIAL: NCT06389006
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of Disitamab Vedotin Combined With Toripalimab Sequential Chemotherapy as Neoadjuvant Treatment in Patients With HR-positive, HER2-low Breast Cancer
Brief Title: To Evaluate the Efficacy and Safety of Disitamab Vedotin Combined With Toripalimab Sequential Chemotherapy as Neoadjuvant Treatment in Patients With HR-positive, HER2-low Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C025
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HR-positive; HER2 low-expressing
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; Injections; toripalimab; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin combined with Toripalimab sequential chemotherapy（Epirubicin +CTX） (Experimental): Disitamab Vedotin combined with Toripalimab sequential chemotherapy arm
  Interventions: Drug: Disitamab Vedotin for Injection; Drug: Toripalimab; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Disitamab Vedotin for Injection — 2.0mg/kg, intravenous infusion，D1, every 2 weeks, Every 6 weeks is a treatment cycle. A total of 2 cycles (12 weeks) of treatment are performed
  Other Names: RC48
Drug: Toripalimab — 3.0 mg/kg, intravenous infusion, D1, every 2 weeks, every 6 weeks is a treatment cycle. A total of 2 cycles (12 weeks) of treatment are performed. Sequential therapy 3.0 mg/kg, intravenous infusion, D1, every 2 weeks,every 6 weeks is a treatment cycle. A total of 2 cycles (12 weeks) of treatment are performed.
  Other Names: JS001
Drug: Epirubicin — According to body surface area, 90mg/m2, intravenous infusion, D1, every 3 weeks, Every 6 weeks is a treatment cycle. A total of 12 weeks of treatment are performed.
Drug: Cyclophosphamide — According to body surface area,600mg/m2, intravenous infusion, D1, every 3 weeks , Every 6 weeks is a treatment cycle. A total of 12 weeks of treatment are performed
  Other Names: CTX

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Disitamab Vedotin combined with Toripalimab sequential chemotherapy as in patients with HR-positive, HER2-low breast cancer

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter phase II clinical trial to evaluate the efficacy and safety of Disitamab Vedotin combined with Toripalimab sequential chemotherapy as neoadjuvant treatment in patients with HR-positive, HER2-low breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign the informed consent;
2. Age ≥18 years old (including the threshold value);
3. Histologically confirmed invasive breast cancer with clinical stage T1c-T2(≥2cm)cN1-2M0 or T3cN0-2M0;
4. As assessed by the research Center, the subjects can tolerate and plan to undergo radical surgery for breast cancer and have not previously received any anti-tumor systemic therapy for breast cancer;
5. Invasive breast tumor tissue with low HER2 expression confirmed by the central laboratory is defined as IHC 1+ or IHC 2+ expression of HER2 protein detected by immunohistochemistry (IHC), and no amplification detected by in situ hybridization (ISH) (according to the Breast Cancer HER2 Detection Guidelines 2019); Primary tumor specimens (wax pieces, slices or fresh tissues) can be provided for HER2 detection;
6. According to the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) 2020 guidelines, tumor tissue estrogen receptor (ER) and progesterone receptor (PgR) expression ≥ 1%;
7. Histological grade (Nottingham grading system) G3 or G2 with ER expression
8. ECOG physical status 0 or 1;
9. At least one measurable lesion according to RECIST v1.1 standard;
10. Heart function:

    1. New York Heart Association (NYHA) Grade < 3;
    2. left ventricular ejection fraction ≥50%;
11. Bone marrow or organ function should meet the following criteria within 7 days before the study dose:

    Hemoglobin ≥ 90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet ≥ 100 ×109/L; Serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); Aspartate aminotransferase (AST) and glutamic pyruvic transaminase (ALT) ≤ 2.5 times the upper limit of normal value; International normalized ratio (INR) and activated partial thrombin time ≤ 1.5×ULN; Serum creatinine ≤ 1.5×ULN or creatinine clearance (CrCl) ≥ 50 mL/min according to Cockcroft-Gault formula method;
12. Fertile female subjects who meet the following conditions

    1. A serum pregnancy test (minimum sensitivity 25 mIU/mL or equivalent units of β-human chorionic gonadotropin [β-hCG]) must be negative within 72 hours before the first dosing of the study intervention. Subjects with false positive results who are confirmed not to be pregnant are eligible for study.
    2. Must agree to contraception for the duration of the study and for at least 6 months after the last dose of investigational drug.
    3. Must agree not to breastfeed or donate eggs from the time of signing the informed consent until 6 months after the last dose of investigational drug.
    4. If sexually active and likely to result in pregnancy, continuous use of at least 2 acceptable forms of contraception, at least 1 of which must be highly effective from the time of the informed consent and continue until at least 6 months after the last dosing of the investigational drug.
13. Fertile male subjects who meet the following conditions

    1. Must agree not to donate sperm from the time of signing the informed consent until at least 4 months after the last dose of investigational drug.
    2. If sexual activity with a fertile person is likely to result in pregnancy, continuous use of at least 2 acceptable forms of contraception, at least 1 of which must be highly effective from the time of the informed consent and continue until at least 4 months after the last dosing of the investigational drug.
    3. If sexually active with a pregnant or breastfeeding patient, condom use must continue from informed consent until at least 4 months after the last dosing of the investigational drug.
14. Able to understand trial requirements, willing and able to follow trial and follow-up procedures.

Exclusion Criteria:

1. Bilateral invasive breast cancer;
2. Previous history of invasive breast cancer;
3. Previously had carcinoma in situ of the breast and received adjuvant endocrine therapy within 5 years of surgery;
4. Use of the investigational drug or major surgery within 4 weeks prior to study dosing;
5. Have received or plan to receive live or attenuated vaccine within 4 weeks before the start of study dose;
6. Previous history of receiving allogeneic hematopoietic stem cell transplantation or organ transplantation;
7. Previous treatment with PD-(L)1, PD-L2, CTLA4 inhibitors and other Antibody-Drug Conjugates;
8. Uncontrolled or significant cardiovascular and cerebrovascular diseases
9. Presence of other treatable or serious lung diseases, including but not limited to active tuberculosis, interstitial lung disease, etc.;
10. Suffering from an active infection that requires systematic treatment;
11. Have active autoimmune diseases requiring systemic treatment within the past 2 years, allowing for relevant replacement therapy;
12. Have a clear past or present history of neurological or psychiatric disorders, including epilepsy or dementia;
13. Persistent ≥ grade 2 sensory or motor neuropathy;
14. In the judgment of the investigator, there is a serious concomitant disease that endangers the safety of the subject or interferes with the completion of the clinical study;
15. Positive HIV test result; Patients with active hepatitis B or C; Persistent coronavirus (COVID-19) infection;
16. Known hypersensitivity or delayed anaphylaxis to certain components of Disitamab Vedotin, and Toripalimab or Certain components of chemotherapy drugs or similar drugs used in the study;
17. Suffering from another malignancy within 5 years prior to signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR) rate | 1month after surgery
  Defined as the proportion of participants with a pathological assessment of pCR (ypT0/Tis, ypN0) in the analyzed population

SECONDARY OUTCOMES:
Breast pathological complete response（bpCR） | 1 month after surgery
  Defined as the proportion of participants with a pathological assessment of bpCR in the analyzed population
Event free survival (EFS) | Up to approximately 3 or 5 years
  The time from random assignment to disease progression, including local progression before surgery; disease recurrence-local, regional, distant, ipsilateral noninvasive, or contralateral (invasive or noninvasive)-or death from any cause
Disease-free survival (DFS) | Up to approximately 3 or 5 years
  From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause including 3- and 5-year event-free survival
Objective Response Rate (ORR) | Baseline to surgery
  Objective response rate.ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
Adverse events (AEs) | Up to approximately 2 months after surgery
  To evaluate safety including adverse event rate and adverse event grade
Change in cluster of differentiation 8 (CD8) | At baseline to surgery
  CD8 in tumor samples by biopsy at baseline and by surgery immediately after surgery would be evaluated by HE or immune staining.
Health-related quality of life - EORTC-QLQ-C30 | Up to approximately 2 years
  Change from baseline in the physical functioning subscale of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden
Residual cancer burden score | 1 month after surgery
  According to the extent of the residual cancer in the primary breast cancer site (mm*mm), the residual cancer (mm*mm), cell density of residual cancer (%), proportion of carcinoma in situ (%), number of positive lymph nodes and maximum diameter of lymph node metastasis (mm), the RCB index and corresponding RCB classification can be obtained. The RCB index and the corresponding RCB grade can be obtained based on the maximum diameter of the cancer (mm).
Change in tumor-infiltrating lymphocytes (TILs) | At baseline to surgery
  Defined as infiltrating lymphocytes isolated from tumor tissue.TILs in tumor samples by biopsy right before the first neoadjuvant therapy (baseline) and by surgery immediately after surgery would be evaluated by HE or immune staining.
Change in programmed cell death protein L1 (PD-L1) | At baseline to surgery
  PD1 in tumor samples by biopsy at baseline and by surgery immediately after surgery would be evaluated by HE or immune staining.

CONTACTS AND LOCATIONS:
Overall Officials: Leng Kang, Study Director — RemeGen Co., Ltd.
Locations (1):
- Jiong Wu, Shanghai, Fudan University Shanghai Cancer Center, China

IPD SHARING:
Plan to Share IPD: No